CLINICAL TRIAL: NCT05470530
Title: Dexamethasone Intravenous Versus Intrathecal in Prolonging the Duration of Spinal Anesthesia and Postoperative Analgesia in Elective Cesarean Section
Brief Title: Dexamethasone Intravenous Versus Intrathecal in Spinal Anesthesia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Marwa Emam, Lecturer, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FMASU MS 179/2022
Record Dates: First submitted 2022-07-20; First posted 2022-07-22 (Actual); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Healthy
Keywords: Dexamethasone, spinal anesthesia, cesarean section
MeSH Terms: interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IT group (Active Comparator): Participants were received normal saline 2 mL intravenously with intrathecal injection of heavy bupivacaine 0.5% 2 mL (10mg) plus 0.5 mL (2mg) dexamethasone diluted in 0.5 ml of 0.9% saline, overall 3 ml volume intrathecally. The dose of 2mg of dexamethasone was demonstrated by Amer (2018) to be the least effective intrathecal dose.
  Interventions: Drug: Dexamethasone
- IV group (Active Comparator): Participants were received dexamethasone 2 mL (8mg) intravenously with intrathecal injection of heavy bupivacaine 0.5% 2 mL plus 1 mL of 0.9% saline
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Dexamethasone — Dexamethasone was given either intrathecal or intravenous in spinal anesthesia during ceaseran section while normal saline was given in control group

SUMMARY:
The purpose of this study is to compare the the effect of intravenous and the intrathecal dexamethasone when added to spinal anesthesia in cesarean section.

DETAILED DESCRIPTION:
1. Pre-operative settings:

   Detailed preoperative examination and preoperative investigations (complete blood picture, Bleeding Time, prothrombin time and partial thromboplastin time) were performed. Age and weight were recorded. The patient was fasting for 8 hours preoperatively.

   In the preanesthetic room, 18-gauge intravenous cannula was sited. Patients was preloaded with 5 mL/kg of lactated Ringer's solution over 20 minutes. The visual analogue scale (VAS) for pain was explained to the patients
2. Intra-operative Settings Inside the operating room, mean arterial blood pressure (MAP), heart rate (HR), electrocardiography (ECG) and peripheral oxygen saturation (SpO2) were obtained using standard non-invasive monitors and base line values were recorded.

The spinal technique was performed under complete aseptic condition with the patient in sitting position at the L3- L4 or L4 -L5 intervertebral space with 25-gauge spinal needle through midline approach. The spinal drugs were administered over 30 second according to each group.

Groups:

The eligible patients were enrolled in this double blinded study and randomly allocated to one of three groups by computer generated random number lists. The allocation was concealed using closed opaque envelopes. The solution for intrathecal injection was prepared by an anesthesiologist who did not have a further role in the study.

Control group (n= 22): Participants were received normal saline 2 mL intravenously with intrathecal injection of heavy bupivacaine 0.5% 2 mL (10mg) plus 1 mL of 0.9% saline, overall 3 ml volume intrathecally (Pyasetska, 2020).

IT group (n= 22): Participants were received normal saline 2 mL intravenously with intrathecal injection of heavy bupivacaine 0.5% 2 mL (10mg) plus 0.5 mL (2mg) dexamethasone diluted in 0.5 ml of 0.9% saline, overall 3 ml volume intrathecally. The dose of 2mg of dexamethasone was demonstrated by Amer (2018) to be the least effective intrathecal dose.

IV group (n= 22): Participants were received dexamethasone 2 mL (8mg) intravenously with intrathecal injection of heavy bupivacaine 0.5% 2 mL plus 1 mL of 0.9% saline (Pyasetska, 2020).

After completing the intrathecal injection, the patient was immediately placed in the supine position IV Ringer's solution 10 ml/kg/hour was administered throughout the surgery. Oxygen was administered through a nasal cannula in a rate of 2 L/min.

Measurements:

Sensory block was assessed according to loss of sensation using cold alcohol swab every two minutes after completing the spinal injection. Time to reach the sensory level of T10 was recorded to determine the effect of the drug on the onset of the spinal anesthesia.

Spinal anesthesia was considered adequate to undergo surgery if the sensory level reaches a T4 level, otherwise the patients were excluded from the study, recorded as "excluded due to low level" and replaced by another patient to achieve the required sample size.

The highest level reached within 30 min, and its time, were recorded. Hemodynamic parameters (heart rate and mean arterial pressure) and SpO2 were measured and recorded just after performing spinal anesthesia, and at 10 min interval till the end of the surgery.

Bradycardia, defined as a heart rate decrease more than 20% of the baseline (preoperative) value, will be treated by atropine 0.6 mg IV.

Hypotension, defined as a decrease in MAP more than 20% of the baseline value, will be treated by IV ephedrine 3 mg IV increments.

Episodes of bradycardia and hypotension and doses of administered drugs for treatment were recorded.

A decrease of SpO2 below 92% was treated by increasing the oxygen flow rate and management of the airway if necessary. The occurrence of this event was recorded.

Occurrence of side effects as nausea, vomiting, itching or shivering were recorded.

Time to two-segment regression of the sensory block from the highest level. The level was assessed every 10 minutes, after reaching the highest sensory level, by loss of sensation to cold alcohol swab. This time was considered as the duration of the sensory block

ELIGIBILITY:
Inclusion Criteria:

* Female patients in childbearing period with an age of 18 years up to 40 years old scheduled to undergo elective cesarean section under spinal anesthesia.

All patients were of ASA II physical status with uncomplicated pregnancy and no comorbidity.

Exclusion Criteria:

* Refusal of procedure or participation in the study by patients. Emergency cesarean section. Any contraindication to spinal anesthesia as infection at site of injection or history or evidence of coagulopathy.

Congenital anomaly of the spine. Psychiatric illness affecting the ability to properly communicate with the patient or to use the VAS for pain.

Receiving analgesics or corticosteroid drugs. Allergies to drugs used.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2022-03-10 (Actual); Primary Completion 2022-07-10 (Actual); Study Completion 2022-07-15 (Actual)

PRIMARY OUTCOMES:
Duration of sensory block in spinal anesthesia | 4 months after starting the study
  The primary objective of this study is to compare the efficacy of intrathecal dexamethasone with dexamethasone when used intravenously as an adjuvant to prolong the sensory block obtained by spinal anaesthesia and postoperative analgesia in cesarean section

CONTACTS AND LOCATIONS:
Overall Officials: Marwa M Mohamed, Lecturer, Principal Investigator — Ain Shams University
Locations (1):
- Faculty of Medicine Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes